CLINICAL TRIAL: NCT04351243
Title: A Multi-Center, Adaptive, Randomized, Double-blind, Placebo-controlled Study to Assess the Efficacy and Safety of Gimsilumab in Subjects With Lung Injury or Acute Respiratory Distress Syndrome Secondary to COVID-19 (BREATHE)
Brief Title: A Study to Assess the Efficacy and Safety of Gimsilumab in Subjects With Lung Injury or Acute Respiratory Distress Syndrome Secondary to COVID-19 (BREATHE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kinevant Sciences GmbH (Industry)
Collaborators: Roivant Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KIN-1901-2001
Record Dates: First submitted 2020-04-15; First posted 2020-04-17 (Actual); Results first posted 2021-12-10 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
Keywords: Granulocyte macrophage-colony stimulating factor (GM-CSF); Immunomodulator; Cytokine storm; COVID-19; Coronavirus; Severe Acute Respiratory Syndrome (SARS); Lung Injury; Monoclonal antibody
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Coronavirus Infections; Severe Acute Respiratory Syndrome; Lung Injury | interventions — gimsilumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gimsilumab (Experimental): Gimsilumab 400 mg on Day 1 Gimsilumab 200 mg on Day 8
  Interventions: Drug: Gimsilumab
- Placebo (Placebo Comparator): Normal saline on Day 1 Normal saline on Day 8
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gimsilumab — Gimsilumab is a fully human monoclonal antibody (mAb).
  Other Names: KIN-1901
  Arms: Gimsilumab
Drug: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
Study KIN-1901-2001 is a multi-center, adaptive, randomized, double-blind, placebo-controlled study to assess the efficacy and safety of gimsilumab in subjects with lung injury or acute respiratory distress syndrome (ARDS) secondary to COVID-19.

DETAILED DESCRIPTION:
Gimsilumab is a monoclonal antibody against granulocyte macrophage-colony stimulating factor (GM-CSF), which is a myeloid cell growth factor and pro- inflammatory cytokine. Late stages of COVID-19 can be marked by a "cytokine storm" and the overactivation of inflammatory myeloid cells that infiltrate and damage tissue, such as the lungs. Inhibition of GM-CSF may be able to reverse this pathology. The anti-GM-CSF mechanism is distinct from antiviral therapeutic mechanisms and may provide synergistic effects when used in combination.

Study KIN-1901-2001 will consist of a 2-week treatment period (last dose Day 8, if administered) and a 22-week follow-up period, for a total study duration of 24 weeks for each subject. A total of 270 subjects (135 subjects per arm) who have a confirmed diagnosis of COVID-19 with clinical evidence of acute lung injury or ARDS will be entered into the trial.

Subjects will receive a 400 mg dose of gimsilumab on Day 1 and a 200 mg dose of gimsilumab on Day 8, or matching placebo (saline solution) on Day 1 and on Day 8. The Day 8 dose will be omitted if the subject is discharged from the hospital prior to the dose or is no longer in need of supplemental oxygen or ventilatory support for >48 hours.

The primary objective of Study KIN-1901-2001 is to evaluate the impact of IV treatment with gimsilumab on mortality in subjects with lung injury or ARDS secondary to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female age ≥18 years, inclusive
2. Subject (or legally authorized representative) is able and willing to provide written informed consent, which includes compliance with study requirements and restrictions listed in the consent form
3. Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR or other approved clinical testing prior to randomization
4. Radiographic evidence of bilateral infiltrates
5. Subject requires high-flow oxygen or meets clinical classification for ARDS
6. Elevated serum CRP or ferritin
7. Subjects who have been treated with convalescent plasma (CP) prior to enrollment are eligible if the subject continues to meet all inclusion criteria at screening
8. The use of investigational anti-viral treatment (e.g., remdesivir) is allowed if the subject continues to meet all inclusion criteria at screening

Additional inclusion criteria are detailed in the protocol

Exclusion Criteria:

1. Evidence of life-threatening dysrhythmia or cardiac arrest on presentation
2. Intubated >72 hours
3. Absolute neutrophil count < 1,000 per mm3
4. Platelet count < 50,000 per mm3
5. AST or ALT > 5X upper limit of normal
6. eGFR <30 mL/min/1.73m2 or requiring hemofiltration or dialysis
7. History of known anti-GM-CSF autoantibodies or pulmonary alveolar proteinosis
8. Severe chronic respiratory disease (e.g., COPD, PAH, IPF, ILD) requiring supplemental oxygen therapy or mechanical ventilation pre-hospitalization (e.g., prior to COVID-19 diagnosis)
9. Use of any immunomodulatory biologic, cell therapy, or small molecule JAK inhibitor within past 7 days or 5 half lives or planned use of any of these agents unless approved by medical monitor
10. Chronic (>4 weeks) use of corticosteroids >10mg/day of prednisone or equivalent
11. Known or suspected active and untreated TB, HIV, hepatitis B or C infection

Additional exclusion criteria are detailed in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Banner University Medical Center, Phoenix, Arizona
  - HonorHealth John C. Lincoln Medical Center, Phoenix, Arizona
  - HonorHealth Scottsdale Osborn Medical Center, Scottsdale, Arizona
  - HonorHealth, Scottsdale, Arizona
  - HonorHealth Scottsdale Shea Medical Center, Scottsdale, Arizona
  - Banner University Medical Center, Tucson, Arizona
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Miami Cancer institute, Miami, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - NorthShore University HealthSystem, Evanston, Illinois
  - East Jefferson General Hospital, Metairie, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Mount Sinai Beth Israel, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Morningside, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Jack & Jane Hamilton Heart and Vascular Hospital, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Baylor Scott & White All Saints Medical Center, Fort Worth, Texas
  - Memorial Hermann Hospital Affiliated with University of Texas Health Science Center at Houston, McGovern Medical School, Houston, Texas
  - Baylor Scott & White Medical Center, Irving, Texas
  - Baylor Scott & White Heart Hospital, Plano, Texas
  - Baylor Scott & White Medical Center, Plano, Texas
  - Baylor Scott & White Medical Center, Round Rock, Texas
  - Baylor Scott & White Medical Center, Temple, Texas
  - Inova Fairfax Medical Campus, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Criner GJ, Lang FM, Gottlieb RL, Mathews KS, Wang TS, Rice TW, Madduri D, Bellam S, Jeanfreau R, Case AH, Glassberg MK, Lyon GM, Ahmad K, Mendelson R, DiMaio JM, Tran MP, Spak CW, Abbasi JA, Davis SG, Ghamande S, Shen S, Sherman L, Lowry S. Anti-Granulocyte-Macrophage Colony-Stimulating Factor Monoclonal Antibody Gimsilumab for COVID-19 Pneumonia: A Randomized, Double-Blind, Placebo-controlled Trial. Am J Respir Crit Care Med. 2022 Jun 1;205(11):1290-1299. doi: 10.1164/rccm.202108-1859OC. PMID 35290169

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gimsilumab | Placebo
Started | 114 | 113
Completed Baseline Assessment | 113 | 112
Completed | 74 | 75
Not Completed | 40 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gimsilumab | Placebo | Total
Number analyzed (Participants) | 113 | 112 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (14.66) | 60.4 (14.27) | 60.2 (14.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 31 | 71
  Male | 73 | 81 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 59 | 42 | 101
  Not Hispanic or Latino | 54 | 70 | 124
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 5 | 6 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 29 | 45
  White | 61 | 52 | 113
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 30 | 23 | 53

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Mortality
Description: "Incidence" is defined as the percent of subjects that died by Day 43
Time Frame: Day 43
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Groups:
- Gimsilumab: Gimsilumab 400 mg on Day 1 Gimsilumab 200 mg on Day 8 Gimsilumab:Gimsilumab is a fully human monoclonal antibody (mAb)
- Placebo: Normal saline on Day 1 Normal saline on Day 8 Placebo: Normal saline
Arm/Group | Gimsilumab | Placebo
Number analyzed (Participants) | 113 | 112
Participants | 32 | 26
Statistical Analysis 1: Comparison: Gimsilumab vs Placebo; Test type: Superiority; p = 0.1885, Mantel Haenszel — one-sided p value; Risk Difference (RD) = 0.05, 95% CI 2-sided [-0.06 to 0.17]

2. Secondary Outcome: Proportion of Subjects Who Are Alive and Not on Mechanical Ventilation
Time Frame: Day 29
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Gimsilumab | Placebo
Number analyzed (Participants) | 113 | 112
Participants | 80 | 78

3. Secondary Outcome: Number of Ventilator-free Days
Description: Subjects who die will be assigned "0" ventilator-free days
Time Frame: Baseline to Day 29
Population: Intent-to-Treat
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Gimsilumab | Placebo
Number analyzed (Participants) | 113 | 112
Days | 29.0 [2.0 to 29.0] | 29.0 [4.0 to 29.0]

4. Secondary Outcome: Time to Hospital Discharge
Time Frame: Baseline to Day 43
Population: Intent-to-Treat
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Gimsilumab | Placebo
Number analyzed (Participants) | 113 | 112
Days | 13.0 [10.0 to 18.0] | 15.0 [9.0 to 19.0]

ADVERSE EVENTS:
Time Frame: Adverse events through Day 43
Arm/Group | Gimsilumab | Placebo
All-Cause Mortality (participants affected / at risk) | 32/113 | 31/112
Serious Adverse Events (participants affected / at risk) | 47/113 | 45/112
Other Adverse Events (participants affected / at risk) | 84/113 | 77/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gimsilumab (N=113) | Placebo (N=112)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 20 (21)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 6 (6)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 8 (8) | 2 (2)
Death (General disorders) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 5 (5) | 0 (0)
Septic shock (Infections and infestations) | 7 (7) | 6 (6)
Pneumonia pseudomonal (Infections and infestations) | 2 (2) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 3 (3)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Viral sepsis (Infections and infestations) | 1 (1) | 0 (0)
Candida sepsis (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Severe acute respiratory syndrom (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Complications associated with device (General disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3) | 9 (9)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 3 (3)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 3 (3)
Venous thrombosis limb (Vascular disorders) | 2 (2) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 4 (4)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 2 (2)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Blood loss anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Intensive care unit acquired weakness (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gimsilumab (N=113) | Placebo (N=112)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 21 (22) | 20 (22)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 6 (6)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6)
Septic shock (Infections and infestations) | 8 (8) | 8 (8)
Pneumonia (Infections and infestations) | 7 (7) | 3 (3)
Sepsis (Infections and infestations) | 6 (6) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 9 (9) | 8 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 5 (5)
Hypernatraemia (Metabolism and nutrition disorders) | 3 (3) | 6 (6)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 8 (9)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 6 (7)
Leukocytosis (Blood and lymphatic system disorders) | 6 (6) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 11 (12) | 14 (14)
Constipation (Gastrointestinal disorders) | 10 (10) | 8 (8)
Hypotension (Vascular disorders) | 8 (8) | 9 (10)
Shock (Vascular disorders) | 1 (1) | 6 (6)
Multiple organ dysfunction syndrome (General disorders) | 9 (9) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 8 (8) | 6 (6)

LIMITATIONS AND CAVEATS:
The Sponsor stopped enrollment of subjects prior to achieving the planned sample size of 270. At the completion of study enrollment, 227 subjects were randomized and 225 received at least one dose of gimsilumab or placebo. All randomized subjects (227 subjects), where possible, completed all study-related activities and had data collected through the planned Day 43 and Day 169 analyses. No safety findings were observed which warranted study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PIs generally may not publish/present on study results before sponsor's first publication. If there is no sponsor publication within 12-18 months after study completion [timeframe may vary among PIs], PIs may publish/present results from only their site, provided the PI submits the publication to sponsor for review. Upon sponsor's request, PIs must delete references to sponsor's confidential information and delay publication to allow sponsor to obtain IP protection.

DOCUMENTS (2):
  • Study Protocol (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT04351243/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/43/NCT04351243/SAP_001.pdf